CLINICAL TRIAL: NCT01812291
Title: Efficacy of a Stepped Care Approach to Manage Depression in Diabetic Patients and Putative Inflammatory Mechanisms Between Diabetes and Depression
Brief Title: Evaluation of a Stepped Care Approach to Manage Depression in Diabetes
Acronym: Ecce_homo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Diabetes Center (Other); Heinrich-Heine University, Duesseldorf (Other); University of Giessen (Other); Helmholtz Zentrum München (Industry); Coordination Center for Clinical Trials (KKS) (Unknown)
Responsible Party: Principal Investigator, Norbert Hermanns, PhD, Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKZ 01GI1107
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder; Minor Depressive Disorder; Sub-Threshold Depression; Diabetes Mellitus
Keywords: Major Depression; Minor Depression; Sub-Threshold Depression; Affective Condition; Mood Disorder; Light Affective Disorder; Subclinical Depressive Symptoms; Diabetes Mellitus; Diabetes-Related Distress; Self-Care Behaviour; Glycaemic Control; Inflammatory Markers
MeSH Terms: conditions — Depressive Disorder, Major; Diabetes Mellitus; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped Care Approach for Depression (Experimental): Step 1: Diabetes-Specific CBT (5 group sessions)
  Step 2: Depression-Specific CBT (6 single sessions)
  Step 3: Referral to Psychotherapist and/or Psychiatrist
  Interventions: Behavioral: Step 1: Diabetes-Specific CBT (5 group sessions); Behavioral: Step 2: Depression-Specific CBT (6 single sessions); Behavioral: Step 3: Referral to Psychotherapist and/or Psychiatrist
- Treatment-as-usual (Active Comparator): Standard Diabetes Education
  Interventions: Behavioral: Standard Diabetes Education

INTERVENTIONS:
Behavioral: Step 1: Diabetes-Specific CBT (5 group sessions) — Diabetes-Specific CBT (5 group sessions) focusing on diabetes-related problems and distress ('DIAMOS - Strengthening Diabetes Motivation').
  Includes:
  * Diabetes problem analysis/ definition
  * Diabetes problem solving intervention
  * Cognitive restructuring of diabetes problems
  * Activation of personal and social resources
  * Goal definition and agreement
  Arms: Stepped Care Approach for Depression
Behavioral: Step 2: Depression-Specific CBT (6 single sessions) — Depression-Specific CBT (6 single sessions) focusing on depressive cognitions and affective problems (manualised).
  Includes:
  * Functional explanatory model of depression
  * Cognitive restructuring of negative thoughts
  * Practice of alternative beneficial thoughts
  * Specific cognitive interventions regarding self-criticism, guilt, low self-esteem, fear, and inactivity.
  Arms: Stepped Care Approach for Depression
Behavioral: Step 3: Referral to Psychotherapist and/or Psychiatrist — Non-responders to previous treatment steps will be referred to an psychotherapist and/or psychiatrist for intensified treatment. Treatments procedures will be monitored and interventions will be scored to enable the evaluation of treatment effects.
  Arms: Stepped Care Approach for Depression
Behavioral: Standard Diabetes Education — Standard diabetes education and professional care.
  Includes:
  * Health care and specific topics (e. g. blood pressure)
  * Diabetes complications
  * Healthy and unhealthy foods, cooking recommendations and recipes
  * Foot care: exercises, care and control, injuries, and diabetic neuropathy
  * Sports, activities and exercise
  * Social aspects of living with diabetes
  Arms: Treatment-as-usual

SUMMARY:
The study examines the efficacy of a stepped care approach for depressed diabetes patients (first study objective). 256 patients with diabetes and comorbid subthreshold or clinical depression will be randomly assigned to either a stepped care approach or a treatment-as-usual condition. The stepped care approach consists of three treatment steps comprising diabetes-specific cognitive-behavioral therapy (CBT) (group), depression-specific CBT (single), and psychotherapeutic and/or psychiatric treatment (single). Patients assigned to the stepped care approach will be treated stepwise until a clinically significant reduction of depressive symptoms is attained or all three treatment steps are passed.

The primary outcome of the first study objective is a clinically significant reduction of depressive symptoms in the 12-month follow-up. Secondary outcomes are reduction of diabetes-related distress and improvement of well-being, health-related quality of life, diabetes acceptance, diabetes self-care, and glycaemic control. Additionally, cost-benefit analyses will be performed.

The second study objective is to analyse associations between diabetes, depression, and the serum levels of inflammatory markers.

The third study objective is to analyse the courses of depressive conditions in diabetes with regard to recovery rates and incidence of major depression.

DETAILED DESCRIPTION:
Compared to persons without diabetes, rates of depressive disorders and mood are doubled in diabetes patients. Epidemiologic studies have shown point prevalence rates of 10 - 14% for major depressive disorder and an additional proportion of almost 20% with subthreshold depression (defined as elevated depressive symptoms without meeting criteria for a specified clinical disorder). Depression and subthreshold depression in diabetes are associated with reduced quality of life, increased diabetes-related distress, and elevated health care costs. Furthermore, depression as well as subthreshold depression seem to be major barriers to an effective self-management of the disease and have been associated with reduced glycaemic control and hyperglycaemia. Both conditions seem to be independent prognostic factors for subsequent morbidity and mortality in diabetes.

Depressive conditions are commonly treated with psychotherapeutic or pharmacologic antidepressive therapies. Since the majority of diabetes patients is suffering from subthreshold depression, evaluated and suitable specific intervention concepts are rare. Moreover, the large variation of symptom levels of depressive patient groups suggests that different types of treatment with different treatment intensities may be required to match individual demands. The issue of 'optimal' treatment also regards concerns about overtreatment and undertreatment of particular patient groups with depressive conditions. Thus, an successive order of treatment steps of increasing intensity appears useful. Since depression in diabetes often is associated with high diabetes-related problems and distress, diabetes-specific as well as depression-specific interventions may be required.

We developed a stepped care approach with three treatment steps comprising diabetes-specific CBT (group), depression-specific CBT (single), and psychotherapeutic and/or psychiatric treatment (single).

The study is a randomized efficacy trial in which the efficacy of the stepped care approach is compared to a treatment-as-usual condition (standard diabetes education). 256 patients with diabetes and comorbid subthreshold or clinical depression will be randomly assigned to either the stepped care approach or the treatment-as-usual condition. Patients assigned to the stepped care approach will be treated stepwise until a clinically significant reduction of depressive symptoms is attained or all three treatment steps are passed.

The primary outcome is a clinically significant reduction of depressive symptoms in the 12-month follow-up. Secondary outcomes are reduction of diabetes-related distress and improvement of well-being, health-related quality of life, diabetes acceptance, diabetes self-care, and glycaemic control. The decisive measurement of this outcomes are conducted 12 months after the treatment (12 month follow up). Additionally, cost-benefit analyses will be performed.

Besides testing the efficacy of the stepped care approach (first objective), there are two additional study objectives:

The second study objective is to analyse associations between diabetes, depression, and the serum levels of inflammatory markers (C-reactive protein (CRP), Interleukin (IL)-6, IL-18, IL-1Ra, Adiponectin, Monocyte chemoattractant protein (MCP)-1). Additionally, the impact of depression treatment on the levels of these markers will be examined.

The third study objective is to analyse the courses of depressive conditions in diabetes with regard to recovery rates and incidence of major depression in subclinically or clinically depressed diabetes patients treated as usual vs. given an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 and <=70
* Diabetes mellitus
* Elevated depressive symptoms (CES-D score >=16) and/or elevated diabetes-related distress (PAID score >=40)
* Sufficient language skills (German)
* Written informed consent

Exclusion Criteria:

* Severe depressive episode (F32.2/ F32.3)
* Current psychotherapeutic/ psychiatric treatment
* Current antidepressive medication
* Suicidal intention
* Current schizophrenia/ psychotic disorder, specified eating disorder, bipolar disorder, addictive disorder, personality disorder
* Severe physical illness (i.e. cancer, multiple sclerosis, dementia)
* Terminal illness
* Bedriddenness
* Guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Depressive Mood - Hamilton Rating Scale for Depression (HAMD) | 12 month
  Mean difference between HAMD scores at baseline and at 12 month follow up

SECONDARY OUTCOMES:
Diabetes-Related Distress - The Problem Areas in Diabetes Questionnaire (PAID) | 12 months
  Mean difference between PAID scores at baseline and at 12 month follow up
Psychological/ Emotional Well-Being - The WHO-5 Well-being Index (WHO-5) | 12 month
  Mean difference between WHO-5 scores at baseline and at 12 month follow up
Health-Related Quality of Life - The Short Form-36 Health Survey (SF-36) | 12 month
  Mean difference between SF-36 scores at baseline and at 12 month follow up
Diabetes Self-Care Behavior - The Summary of Diabetes Self-Care Activities Measure (SDSCA) | 12 month
  Mean differences between SDSCA scores at baseline and at 12 month follow
Glycaemic Control (HbA1c) | 12 month
  Mean differences between HbA1c values at baseline and at 12 month follow
Health-Related Quality of Life - The EuroQol-5D (EQ-5D) | 12 month
  Mean differences between EQ-5D scores at baseline and at 12 month follow
Diabetes Self-Care Behavior - The Diabetes Self-Management Questionnaire (DSMQ) | 12 month
  Mean differences between DSMQ scores at baseline and at 12 month follow

OTHER OUTCOMES:
Inflammatory Markers | Baseline, 12 month follow up
  Serum levels of the inflammatory markers CRP, IL-6, IL-18, IL-1Ra, Adiponectin, MCP-1 are assessed to enable analyses with regard to the second study objective - associations between diabetes, depression, and inflammation. The measurement of this additional outcome variable is conducted twice, at baseline and 12 months after the treatment (12 month follow up).
Major Depressive Disorder | 12 months
  Difference in rates of major depression according to ICD-10 criteria between baseline and 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Kulzer, PD Dr., Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim; Norbert Hermanns, Prof. Dr., Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim; Thomas Haak, Prof. Dr., Study Director — Forschungsinstitut der Diabetes Akademie Mergentheim; Johannes Kruse, Prof. Dr., Principal Investigator — University of Giessen
Locations (1):
- Forschungsinstitut der Diabetes Akademie Mergentheim e. V., Bad Mergentheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Schmitt A, Kulzer B, Ehrmann D, Haak T, Hermanns N. Diabetes Distress and Depression during COVID-19: Response to Breznoscakova et al. Uncovering the Untold Emotional Toll of Living with Diabetes in the COVID-19 Era. Psychother Psychosom. 2022;91(4):288-289. doi: 10.1159/000524602. Epub 2022 May 6. No abstract available. PMID 35526518
- [Result] Schmitt A, Kulzer B, Reimer A, Herder C, Roden M, Haak T, Hermanns N. Evaluation of a Stepped Care Approach to Manage Depression and Diabetes Distress in Patients with Type 1 Diabetes and Type 2 Diabetes: Results of a Randomized Controlled Trial (ECCE HOMO Study). Psychother Psychosom. 2022;91(2):107-122. doi: 10.1159/000520319. Epub 2021 Dec 7. PMID 34875666
- [Result] Herder C, Schmitt A, Budden F, Reimer A, Kulzer B, Roden M, Haak T, Hermanns N. Association between pro- and anti-inflammatory cytokines and depressive symptoms in patients with diabetes-potential differences by diabetes type and depression scores. Transl Psychiatry. 2018 Mar 9;7(11):1. doi: 10.1038/s41398-017-0009-2. PMID 29520075
- [Result] Herder C, Schmitt A, Budden F, Reimer A, Kulzer B, Roden M, Haak T, Hermanns N. Longitudinal associations between biomarkers of inflammation and changes in depressive symptoms in patients with type 1 and type 2 diabetes. Psychoneuroendocrinology. 2018 May;91:216-225. doi: 10.1016/j.psyneuen.2018.02.032. Epub 2018 Mar 6. PMID 29525039
- [Derived] Schmitt A, Reimer A, Kulzer B, Haak T, Gahr A, Hermanns N. Assessment of diabetes acceptance can help identify patients with ineffective diabetes self-care and poor diabetes control. Diabet Med. 2014 Nov;31(11):1446-51. doi: 10.1111/dme.12553. Epub 2014 Aug 2. PMID 25047992